CLINICAL TRIAL: NCT01763450
Title: LIAONING CANCER HOSPITAL&INSTITUTE
Brief Title: Bevacizumab Therapy Untreated Unresectable Liver Metastases From Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Chun Song, Professor, Liaoning Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Avastin Study
Record Dates: First submitted 2012-12-28; First posted 2013-01-08 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2012-09

CONDITIONS: Liver Metastases; Colorectal Cancer
Keywords: Bevacizumab; conversion therapy; liver metastases; colorectal cancer; objective response rate
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab plus chemotherapy (Experimental): 1. Bevacizumab:
     7.5mg/kg, iv, on day 1 of each 21 day cycle or 5mg/kg, iv, on day 1 of each 14 day cycle;
  2. Oxaliplatin+capecitabine(XELOX):( The total dose not less than 70% of the recommended dose of this standard) Oxaliplatin: 130mg/m2,d1; capecitabine: 850-1,000mg/m2，d1-d14, bid，each 21 day cycle;
  3. Oxaliplatin+5-Fluorouracil+ Levomisole（FOLFOX）:
  Oxaliplatin: 85mg/m2,iv for 2 hours ,d1; Levomisole（LV）: 400mg/m2,iv for 2 hours,d1; 5-Fluorouracil（5-FU） :400mg/m2 iv,d1,then 1200mg/m2/d ×2d continuous intravenous infusion(volume dose:2400mg/m2,iv for 46-48 hours ) each 14 day cycle;
  Interventions: Drug: bevacizumab plus chemotherapy

INTERVENTIONS:
Drug: bevacizumab plus chemotherapy — 1. Bevacizumab:
     7.5mg/kg, iv, on day 1 of each 21 day cycle or 5mg/kg, iv, on day 1 of each 14 day cycle;
  2. Oxaliplatin+capecitabine(XELOX):( The total dose not less than 70% of the recommended dose of this standard) Oxaliplatin: 130mg/m2,d1; capecitabine: 850-1,000mg/m2，d1-d14, bid，each 21 day cycle;
  3. Oxaliplatin+5-Fluorouracil+ Levomisole（FOLFOX）:
  Oxaliplatin: 85mg/m2,iv for 2 hours ,d1; Levomisole（LV）: 400mg/m2,iv for 2 hours,d1; 5-Fluorouracil（5-FU） :400mg/m2 iv,d1,then 1200mg/m2/d ×2d continuous intravenous infusion(volume dose:2400mg/m2,iv for 46-48 hours ) each 14 day cycle;

SUMMARY:
A multi-center, non-random, open study ,to observe efficacy and safety of bevacizumab plus Oxaliplatin based multidrug chemotherapy as conversion therapy for patients with previously untreated unresectable liver metastases from colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES：To assess the objective response rate(ORR)（8 weeks after chemotherapy）

SECONDARY OBJECTIVES：

1. To assess the R0 resection rate of liver metastases（8 weeks after chemotherapy、every three months follow-up 1 time in R0 postoperative 1-2 years、Every six months follow-up 1 time in R0 postoperative 2-5 years）
2. To assess the incidence of adverse events of level 3-4 （Bleeding、Gastrointestinal Perforation、Anastomotic Fistula、Hypertension、Wound Healing Delay）（8 weeks after chemotherapy）

ELIGIBILITY:
Inclusion Criteria:

1. Written inform consent form
2. histologically or cytologically confirmed Colorectal Adenocarcinoma
3. Age≥18 and ≤80 years old
4. Primary colorectal cancer and liver metastases，Liver lesions determined to be unresectable by multidisciplinary team (MDT) （primary lesions surgically removed）
5. Simultaneity or heterochrony metastases
6. Colorectal cancer lesions from anal edge at least 8 cm
7. Within 6 months did not receive any chemotherapy, including targeted therapy
8. One or more measurable lesions, conventional Computed Tomography(CT) scanning measurement diameter at least 20 mm [Response Evaluation Criteria In Solid Tumors(RECIST) standard]
9. Eastern Collaborative Oncology Group(ECOG) 0 or 1
10. Expected lifetime at least for 12 weeks
11. Screening within 7 days， the ability of bone marrow, liver and kidney function reserve enough；Absolute neutrophil count（ANC）≥1.5x109/L; hemoglobin≥9.0g/dl; platelet count≥80 x109/L; Total Bilirubin(TBil)≤1.5 x upper level of normal range(ULN); Alanine Aminotransferase(ALT) and Aspartate Aminotransferase(AST)≤2.5 x ULN(Patients with hepatic metastasis≤5x ULN); alkaline phosphatase≤4 x ULN; serum creatinine≤1.5 x ULN;
12. Women of reproductive age should take effective contraceptive measures;

Exclusion Criteria:

1. Arrhythmia requiring medication（except β- receptor blocking pharmacon and digoxigenin），symptomatic coronary artery disease and myocardial ischemia [myocardial infarction (≤6months before enrollment)]，congestive heart failure [≥New York Heart Association(NYHA)2];
2. History of HIV infection,Chronic hepatitis B or hepatitis C of active phase(high copy virus DNA);
3. Other activated serious infection [>National Cancer Institute-Common Toxicity Criteria(NCI-CTC) 3.0];
4. Any extrahepatic metastases;
5. Seizures requiring medication(such as steroids or antiepileptic therapy);
6. Other malignancies in the past 5 years (except curatively treated basal cell carcinoma of the skin and/or in situ carcinoma of the cervix);
7. Chronic inflammatory bowel disease, intestinal obstruction;
8. Drug abuse and medicine, psychology or social conditions may interfere with patients to participate in research or the results of the evaluation have influence;
9. Known or suspected allergy to any investigational drug in this study;
10. Any unstable condition or is likely to endanger the patient safety and compliance situation;
11. Pregnant or lactating women not using or refusing to use effective non hormonal means of contraception;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-05 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
To assess the objective response rate(ORR) | 8 weeks after chemotherapy

SECONDARY OUTCOMES:
To assess the R0 resection rate of liver metastases | 8 weeks after chemotherapy、every three months follow-up 1 time in R0 postoperative 1-2 years、Every six months follow-up 1 time in R0 postoperative 2-5 years

OTHER OUTCOMES:
To assess the incidence of adverse events of level 3-4 （Bleeding、Gastrointestinal Perforation、Anastomotic Fistula、Hypertension、Wound Healing Delay） | 8 weeks after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Chun Song, Ph.D, Principal Investigator — Professor
Locations (2):
- China (2):
  - Second Affiliated Hosptial of Harbin Medical University, Harbin, Heilongjiang
  - Liaoning Cancer Hospital&Institute, Shenyang, Liaoning